CLINICAL TRIAL: NCT06733896
Title: The Effectiveness of Sternocleidomastoid Muscle Pressure Points in Patients with Cervicogenic Headache
Brief Title: SCM Muscle Released in Patients with Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Hosny M Battesha, associate professor hanan hosny M Battesha, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cervicogenic Headache
Record Dates: First submitted 2024-12-05; First posted 2024-12-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cervicogenic Headache
Keywords: trigger points; sternocleidomastoid; headaches
MeSH Terms: conditions — Post-Traumatic Headache; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: trigger point pressure
- control group (Active Comparator)
  Interventions: Other: neck exercises

INTERVENTIONS:
Other: trigger point pressure — The midpoint of the sternocleidomastoid muscle with abundant nerve distribution and the onset and endpoint of the sternocleidomastoid muscle were used as acupoints, which can relieve localised muscle spasms and promote nerve nutrition.
  Arms: study group
Other: neck exercises — Manual Cervical Traction Technique and others
  Arms: control group

SUMMARY:
Sternocleidomastoid syndrome is often characterized by referred pain in other areas. Like all muscles, the SCM can develop tight, and non-contracting bands called trigger points that can refer pain elsewhere. For the SCM, the trigger point referral areas are the eye and forehead, the back of the head (occiput), front of the neck, cheek, and side of the head. Trigger points can be treated by direct manual massage, dry needling, or platelet-poor plasma injection.

DETAILED DESCRIPTION:
Cervicogenic headache is a specific type of headache that originates from the cervical spine and is typically chronic in nature. Diagnostic criteria for CGH have been established by the International Headache Society (IHS) and are cited extensively in the literature. Diagnosis of CGH through manual examination is a more recent practice. To our knowledge, no systematic review of manual diagnosis of CGH has been performed.

ELIGIBILITY:
Inclusion Criteria:

* History of CGH ≥ 3 months at Baseline 1, ≥5 days of CGH per month
* CGH intensity ≥3 (0-10 scale)
* Cervical spine dysfunction (cervical joint tenderness and/or restricted segmental motion)
* Clear temporal sequence linking the source of CGH to the neck: headache preceded by neck pain, stiffness, movement and/or awkward postures

Exclusion Criteria:

* Other headaches within one year of enrollment (e.g. migraine occurring on >1 day per month in the last year, medication overuse, daily, cluster, temporomandibular joint dysfunction related headaches, sinus, posttraumatic, tumor and glaucoma related, occipital neuralgia, metabolic/toxic/substance abuse related).
* Spinal manipulative therapy, massage or exercise therapy for neck pain or headaches in the previous 3 months. Any other types of care by a licensed provider in the previous month for headaches or neck pain
* Contraindications to study treatments (e.g., inflammatory arthropathies, cervical instability, severe osteoporosis, vertigo, dizziness)
* Daily prescription or nonprescription pain medication; corticosteroid use in previous month
* Cancer in the past five years
* ear problem

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
cervical neck pain | 4 weeks
  visual analogue scale: This pain scale is most commonly used. A person rates their pain on a scale of 0 to 10 or 0 to 5. Zero means "no pain," and 5 or 10 means "the worst possible pain."
  These pain intensity levels may be assessed upon initial treatment, or periodically after treatment.

SECONDARY OUTCOMES:
biodex balance system | 4 weeks
  assessment of posture stability, level eight was selected on the (the most stable level), then the dynamic limit of stability testing mode was selected and then the data of each patient were inserted into the device. The patient was instructed to try to achieve a centered position on the platform by moving their feet, once the platform was programmed to move. Visual feedback was provided on screen, with the cursor moving in relation to the feedback from the patients' feet. Once the cursor had been centered, the platform was kept level beneath the patient's feet while the patient was standing in a comfortable upright position
neck stability index | 4 weeks
  It is patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation, each item scored with a possible 0-5 value with the larger number indicating a higher self-reported disability status. The score on this questionnaire can range from 0-50. In order to calculate a percentage, simply multiply the final value by two

CONTACTS AND LOCATIONS:
Locations (1):
- Umm Al Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34003165/